CLINICAL TRIAL: NCT01074294
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo Controlled Study of the Safety and Efficacy of OPC-34712 as Adjunctive Therapy in the Treatment of Adult Attention Deficit/ Hyperactivity Disorder
Brief Title: Study of the Safety and Efficacy of OPC-34712 as a Complementary Therapy in the Treatment of Adult Attention Deficit/Hyperactivity Disorder
Acronym: STEP-A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 331-08-213
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Inattention; Hyperactivity; Impulsivity; Distractibility; Procrastination; Disorganized; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm; Impulsive Behavior | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase A (Single-blind Prospective Treatment Phase): Placebo + Stimulant (Experimental): Participants received single-blind matching-placebo tablets along with open-label stimulant determined by the investigator, once daily for 5 weeks. Once assigned to a stimulant by the investigator, participants remained on the same stimulant for the duration of the trial. Participants who met eligibility criteria i.e., who received prior treatment for adult ADHD and treatment-naïve participants were included in this arm group. Participants with incomplete response at the end of Phase A (Week 5) entered Phase B and rest of the participants continued to Phase A+.
  Interventions: Drug: Placebo; Drug: Stimulant Therapy
- Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant (Experimental): Participants with incomplete response (with a > 0% and < 30% reduction in ADHD Symptoms Total Score {18 items} between the baseline of Phase A and the end of prospective treatment { Week 5} as measured by the CAARS-O:SV { Conners' Adult ADHD Rating Scale-Observer: Screening Version}, and a CAARS-O:SV ADHD Symptoms Total Score {18 items} of ≥ 24 at Week 5, and a clinical global impression - improvement scale (CGI-I) score of 3 or 4 at Week 5) at the end of Phase A (Week 5), received Brexpiprazole 2 milligram (mg) tablet along with stimulant determined by the investigator, once daily for 6 weeks (up to Week 11).
  Interventions: Drug: OPDC-34712; Drug: Stimulant Therapy
- Phase B (Double-blind Randomization Phase): Placebo + Stimulant (Placebo Comparator): Participants with incomplete response (with a > 0% and < 30% reduction in ADHD Symptoms Total Score {18 items} between the Baseline of Phase A and the end of prospective treatment { Week 5} as measured by the CAARS-O:SV, and a CAARS-O:SV ADHD Symptoms Total Score {18 items} of ≥ 24 at Week 5, and a CGI-I score of 3 or 4 at Week 5) at the end of Phase A (Week 5), received matching-placebo tablets along with stimulant determined by the investigator, once daily for 6 weeks (up to Week 11).
  Interventions: Drug: Placebo; Drug: Stimulant Therapy
- Phase A+ (Single-blind Phase A Responders and Non-responders): Placebo + Stimulant (Experimental): Participants with response (with a ≥ 30% reduction in ADHD Symptoms Total Score {18 items} between Baseline of Phase A and the end of prospective treatment { Week 5} as measured by the CAARS-O:SV, or a CAARS-O:SV ADHD Symptoms Total Score {18 items} of < 24 at Week 5, or a CGI-I score of < 3 at Week 5) and non-response (with deterioration or no change in ADHD symptoms at Week 5) at the end of Phase A (Week 5), received single-blind matching-placebo tablets along with open-label stimulant determined by the investigator, once daily for an additional 6 weeks (up to Week 11).
  Interventions: Drug: Placebo; Drug: Stimulant Therapy

INTERVENTIONS:
Drug: OPDC-34712 — OPDC-34712 tablets, daily, Orally.
  Other Names: Brexpiprazole
  Arms: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant
Drug: Placebo — Matching-placebo tablets, daily, Orally.
  Arms: Phase A (Single-blind Prospective Treatment Phase): Placebo + Stimulant; Phase A+ (Single-blind Phase A Responders and Non-responders): Placebo + Stimulant; Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Drug: Stimulant Therapy — Mixed amphetamine salts or Dexmethylphenidate hydrochloride (HCL) or Methylphenidate HCl or Lisdexamfetamine dimesylate as per standard of care.

SUMMARY:
This study tests the effects of an investigational antipsychotic drug (called OPC-34712) in adults with attention deficit hyperactivity disorder (ADHD) when taken with an approved stimulant medication to explore a possible impact on sleep, quality of life and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 to 55 years of age, inclusive, at the time of informed consent.
* Participants with a primary diagnostic and statistical manual of mental disorders, fourth edition, text revision (DSM-IV-TR) diagnosis of ADHD (including inattentive, hyperactive, and combined subtypes) as confirmed by the Conners' Adult ADHD diagnostic interview (CAADID). Participants may have received prior treatment for adult ADHD, may be currently receiving treatment for adult ADHD at screening, or may be treatment-naive.
* Participants willing to discontinue all prohibited psychotropic medication starting from the time of signing the informed consent and during the study period.

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug.
* Participants with an adequate response, as determined by the investigator, to any stimulant taken for the treatment of adult ADHD after 18 years of age.
* Participants with a clinically significant current Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder.
* Participants who participated in a clinical trial within the last 180 days or who participated in more than two clinical trials within the past year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 740 (Actual)
Dates: Start 2010-03-16 (Actual); Primary Completion 2011-06-20 (Actual); Study Completion 2011-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (35):
- United States (35):
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Irvine, California
  - Pasadena, California
  - San Francisco, California
  - Bradenton, Florida
  - Jacksonville, Florida
  - Maitland, Florida
  - North Miami, Florida
  - Orlando, Florida
  - South Miami, Florida
  - Atlanta, Georgia
  - Smyrna, Georgia
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Rochester Hills, Michigan
  - Saint Charles, Missouri
  - Cherry Hill, New Jersey
  - Willingboro, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Woodstock, Vermont
  - Herndon, Virginia
  - Bellevue, Washington
  - Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 37 sites in United States from 16 Mar 2010 to 20 Jun 2011.
Pre-assignment Details: The study consisted of a screening phase, phase A (5-week single-blind prospective treatment phase), phase A+ (6-week single-blind phase A responders and non-responders), and phase B (6-week double-blind randomization phase). 740 participants were enrolled in Phase A, and 574 completed Phase A. Of these, 235 incomplete responders then randomized in 2: 1 ratio to Phase B and 339 responders and non-responders continued in Phase A+.
Groups:
- Phase A (Single-blind Prospective Treatment Phase): Placebo + Stimulant: Participants received single-blind matching-placebo tablets along with open-label stimulant determined by the investigator, once daily for 5 weeks. Once assigned to a stimulant by the investigator, participants remained on the same stimulant for the duration of the trial. Participants who met eligibility criteria i.e., who received prior treatment for adult attention deficit/hyperactivity disorder (ADHD) and treatment-naïve participants were included in this arm group. Participants with incomplete response at the end of Phase A (Week 5) entered Phase B and rest of the participants continued to Phase A+.
- Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant: Participants with incomplete response (with a > 0% and < 30% reduction in ADHD Symptoms Total Score {18 items} between the Baseline of Phase A and the end of prospective treatment {Week 5} as measured by the CAARS-O:SV {Conners' Adult ADHD Rating Scale-Observer: Screening Version}, and a CAARS-O:SV ADHD Symptoms Total Score {18 items} of ≥ 24 at Week 5, and a clinical global impression - improvement scale (CGI-I) score of 3 or 4 at Week 5) at the end of Phase A (Week 5), received Brexpiprazole 2 milligram (mg) tablet along with stimulant determined by the investigator, once daily for 6 weeks (up to Week 11).
- Phase B (Double-blind Randomization Phase): Placebo + Stimulant: Participants with incomplete response (with a > 0% and < 30% reduction in ADHD Symptoms Total Score {18 items} between the Baseline of Phase A and the end of prospective treatment {Week 5} as measured by the CAARS-O:SV, and a CAARS-O:SV ADHD Symptoms Total Score {18 items} of ≥ 24 at Week 5, and a CGI-I score of 3 or 4 at Week 5) at the end of Phase A (Week 5), received matching-placebo tablets along with stimulant determined by the investigator, once daily for 6 weeks (up to Week 11).
- Phase A+ (Single-blind Phase A Responders and Non-responders): Placebo + Stimulant: Participants with response (with a ≥ 30% reduction in ADHD Symptoms Total Score {18 items} between Baseline of Phase A and the end of prospective treatment {Week 5} as measured by the CAARS-O:SV, or a CAARS-O:SV ADHD Symptoms Total Score {18 items} of < 24 at Week 5, or a CGI-I score of < 3 at Week 5) and non-response (with deterioration or no change in ADHD symptoms at Week 5) at the end of Phase A (Week 5), received single-blind matching-placebo tablets along with open-label stimulant determined by the investigator, once daily for an additional 6 weeks (up to Week 11).
Period: Phase A (Day 1 to Week 5)
Arm/Group | Phase A (Single-blind Prospective Treatment Phase): Placebo + Stimulant | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant | Phase A+ (Single-blind Phase A Responders and Non-responders): Placebo + Stimulant
Started | 740 | 0 | 0 | 0
Analyzed for Safety (Safety Sample consisted of randomized participants who received at least one dose of double-blind investigational medicinal product (IMP) as indicated on the dosing record.) | 733 | 0 | 0 | 0
Completed | 574 | 0 | 0 | 0
Not Completed | 166 | 0 | 0 | 0
Not completed — Lost to Follow-up | 16 | 0 | 0 | 0
Not completed — Adverse Event | 51 | 0 | 0 | 0
Not completed — Protocol specified withdrawal criteria | 47 | 0 | 0 | 0
Not completed — Withdrawn From Participation by the Investigator | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 32 | 0 | 0 | 0
Not completed — Protocol deviation | 10 | 0 | 0 | 0
Not completed — Participants not Dosed | 7 | 0 | 0 | 0
Period: Phase B and Phase A+ (Week 6 to Week 11)
Arm/Group | Phase A (Single-blind Prospective Treatment Phase): Placebo + Stimulant | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant | Phase A+ (Single-blind Phase A Responders and Non-responders): Placebo + Stimulant
Started | 0 | 155 | 80 | 339
Analyzed for Safety (Safety Sample consisted of randomized participants who received at least one dose of double-blind IMP as indicated on the dosing record.) | 0 | 155 | 80 | 235
Completed | 0 | 146 | 70 | 314
Not Completed | 0 | 9 | 10 | 25
Not completed — Lost to Follow-up | 0 | 2 | 2 | 11
Not completed — Adverse Event | 0 | 2 | 3 | 8
Not completed — Protocol-Specified Withdrawal Criteria | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 4
Not completed — Protocol Violation | 0 | 0 | 3 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Sample consisted of all participants who were randomized in Phase B. Phase A+ Sample consisted of all non-randomized participants who were Phase A Responders or Phase A Non-responders, and who continued on Stimulant + single-blind placebo beyond Week 5. As pre-specified in the protocol and statistical analysis plan (SAP) the data is reported for Phase B and Phase A+ participants.
Groups:
- Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant: Participants with incomplete response (with a > 0% and < 30% reduction in ADHD Symptoms Total Score {18 items} between the Baseline of Phase A and the end of prospective treatment {Week 5} as measured by the CAARS-O:SV, and a CAARS-O:SV ADHD Symptoms Total Score {18 items} of ≥ 24 at Week 5, and a CGI-I score of 3 or 4 at Week 5) at the end of Phase A (Week 5), received Brexpiprazole 2 mg tablet along with stimulant determined by the investigator, once daily for 6 weeks (up to Week 11).
- Total: Total of all reporting groups
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant | Phase A+ (Single-blind Phase A Responders and Non-responders): Placebo + Stimulant | Total
Number analyzed (Participants) | 155 | 80 | 339 | 574
Age, Continuous [Mean (Full Range); unit: years] | 36.0 [18.0 to 55.0] | 33.6 [18.0 to 55.0] | 33.6 [18.0 to 55.0] | 34.4 [18.0 to 55.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 38 | 164 | 281
  Male | 76 | 42 | 175 | 293
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 10 | 48 | 77
  Not Hispanic or Latino | 136 | 69 | 288 | 493
  Unknown or Not Reported | 0 | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 4 | 6
  Asian | 3 | 0 | 9 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 10 | 38 | 57
  White | 140 | 65 | 281 | 486
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 7 | 13
CAARS-O:SV ADHD Symptoms Total Score (18 items) [Mean (Full Range); unit: score on a scale] — Conners' Adult Attention-deficit/Hyperactivity Disorder (ADHD) Rating Scale-Observer: Screening Version (CAARS-O:SV) is 30 items scale with 3 subscales: Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Inattentive Symptoms (9 items), DSM- IV Hyperactive/Impulsive Symptoms (9 items), and DSM-IV ADHD Index (12 items). Total ADHD Symptoms Score (18 items) consisted of combined score for inattentive symptoms and hyperactive/impulsive symptoms subscales and is scored on 4-point scale from 0(never) to 3(very frequently) for total score ranging from of 0 to 54, higher scores=worsening. Population: Efficacy Sample consisted of participants in the Randomized Sample who had a Baseline value for Phase B (ie, Week 5) and at least one post-randomization efficacy evaluation for CAARS-O:SV ADHD symptoms Total Score (18 items) in Phase B. Phase A+ Sample- all non-randomized participants who were Phase A Responders or Phase A Non-responders, and continued on Stimulant + single-blind placebo beyond Week 5. Number analyzed is the number of participants with data available for analyses at Baseline.
  score on a scale
    number analyzed (Participants) | 153 | 78 | 339 | 570
    (all) | 32.94 [24.00 to 47.00] | 33.99 [24.00 to 52.00] | 40.1 [30.00 to 54.00] | 35.67 [24.00 to 54.00]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (End of Phase A) in the CAARS-O:SV ADHD Symptoms Total Score (18 Items) to End of Phase B
Description: The CAARS-O:SV is a 30 items scale with 3 subscales: Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) Inattentive Symptoms (9 items), DSM- IV Hyperactive/Impulsive Symptoms (9 items), and DSM-IV ADHD Index (12 items). Total ADHD Symptoms Score (18 items) consisted of the combined score for the inattentive symptoms and hyperactive/impulsive symptoms subscales and is scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) for a total score ranging from of 0 to 54, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The Mixed model repeated measures (MMRM) model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: Efficacy Sample consisted of participants in the Randomized Sample who had a Baseline value for Phase B (ie, Week 5) and at least one post-randomization efficacy evaluation for CAARS-O:SV ADHD symptoms Total Score (18 items) in Phase B. As pre-specified in the protocol and SAP the data is reported only for Phase B participants. Overall number analyzed is the number of participants available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 147 | 69
score on a scale | -9.02 (0.77) | -9.71 (1.06)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.5845, Mixed Models Analysis — The p-value was derived using MMRM method with treatment, trial center, visit week, and treatment by visit week interaction as class effects and Week 5 value as covariate; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [-1.80 to 3.19] — The difference between Least Squares (LS) means derived from the MMRM model. This comparison was tested for statistical significance at a 0.05 (two-sided) significance level

2. Secondary Outcome: Change From Baseline (End of Phase A) in Wender-Reimherr Adult Attention Deficit Disorder Scale (WRAADDS) Total Score to End of Phase B
Description: WRAADDS is used to measure the severity of symptoms in adults with ADHD. This structured interview consists of 28 items in 7 psychopathologic domains, which were rated by a clinical expert on a 0 to 2-point Likert scale. The psychopathologic 7 domains are inattention (6 items), impulsivity (3 items), and hyperactivity (3 items), disorganization (5 items), temper (3 items), affective lability (4 items), and emotional over-reactivity (4 items). The scale rated individual items from 0 to 2 (0=not present, 1=mild, 2=clearly present) and summarized each of the 7 categories on a 0-to-4 scale (0=none, 1=mild, 2=moderate, 3=quite a bit, 4=very much). The WRAADDS total score is defined as sum of all 28 item sub scores (range 0 - 56), higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The analysis of covariance (ANCOVA) method was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 150 | 74
score on a scale | -3.93 (0.42) | -3.84 (0.56)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.8832, ANCOVA — The p-value was derived using ANCOVA model with treatment and trial center as main effects and Week 5 value as covariate; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1.37 to 1.18] — The difference between LS means derived from the ANCOVA model. This comparison was tested for statistical significance at a 0.05 (two-sided) significance level

3. Secondary Outcome: Change From Baseline (End of Phase A) in Sleep Improvement Measured by Insomnia Severity Index (ISI) Total Score to End of Phase B
Description: The ISI is self-report instrument that has been validated specifically for measuring the perceived severity of insomnia. The scale was composed of a total of 7 items based on self-report questionnaire based on several indicators assessing the perceived severity of difficulties initiating sleep, staying asleep, and early morning awakenings, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item was rated on a scale from 0 (none) to 4 (higher score indicating greater impairment/concern). A total score ranging from 0 to 28 was calculated from the sum of the individual item scores, higher scores indicate increased severity of insomnia. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 147 | 69
score on a scale | -1.05 (0.41) | -1.62 (0.56)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.3864, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-0.72 to 1.86] — The difference between LS means derived from the MMRM model. This comparison was tested for statistical significance at a 0.05 (two-sided) significance level

4. Secondary Outcome: Change From Baseline (End of Phase A) in Sleep Improvement Measured by ISI for Item 2 Score (Difficulty Staying Asleep) to End of Phase B
Description: as for outcome 3
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 147 | 69
score on a scale | -0.04 (0.08) | -0.37 (0.10)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.0061, Mixed Models Analysis — The p value was derived using MMRM method with treatment, trial center, visit week, and treatment by visit week interaction as class effects and Week 5 value as covariate; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [0.10 to 0.58] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline (End of Phase A) in the Spatial Working Memory (SWM) Between Errors 4-8 Boxes Test Score as Measured by Cambridge Neuropsychological Test Automated Battery (CANTAB) to End of Phase B
Description: ADHD was measured with the CANTAB. SWM test was one of the tasks of CANTAB, SWM measured the ability to retain spatial information and to manipulate remembered items in working memory. This test was sensitive measure of executive dysfunction. Participants search for colored tokens hidden inside boxes on screen by touching them. The critical instruction was that once token has been found inside box, no token was hidden inside that box again, so participants must not return to box where a token was found. The key measurement of the SWM task is the SWM Between Errors 4-8 Boxes, which measured the total number of times a participant revisits a box in which a token has previously been found is measured for the 4, 6, and 8-box stages. Total scores ranged from 0-153. A lower score indicated better performance. The ANCOVA model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 145 | 72
score on a scale | 0.10 (0.67) | -0.31 (0.90)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.6932, ANCOVA — The p-value was derived from ANCOVA model, with treatment and trial center as main effects and Week 5 value as covariate; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-1.64 to 2.46] — This comparison was tested for statistical significance at a 0.05 (two-sided) significance level

6. Secondary Outcome: Change From Baseline (End of Phase A) in CAARS-O:SV ADHD Symptoms Total Score (18 Items) to Each Time Point in Phase B Other Than Week 11
Description: The CAARS-O:SV is a 30 items scale with 3 subscales DSM-IV Inattentive Symptoms (9 items), DSM-IV Hyperactive/Impulsive Symptoms (9 items), and DSM-IV ADHD Index (12 items). Total ADHD Symptoms Score (18 items) consisted of the combined score for the inattentive symptoms and hyperactive/impulsive symptoms subscales and is scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) for total score ranging from of 0 to 54, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Weeks 6, 7, 8, 9 and 10
Population: Efficacy Sample consisted of participants in the Randomized Sample who had a Baseline value for Phase B (ie, Week 5) and at least one post-randomization efficacy evaluation for CAARS-O:SV ADHD symptoms Total Score (18 items) in Phase B. As pre-specified in the protocol and SAP the data is reported only for Phase B participants. Number analyzed is the number of participants with data available for analyses at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Change at Week 6 | -3.82 (0.49) | -4.62 (0.64)
  Change at Week 7: number analyzed (Participants) | 150 | 74
  Change at Week 7 | -5.54 (0.58) | -6.21 (0.78)
  Change at Week 8: number analyzed (Participants) | 150 | 74
  Change at Week 8 | -6.37 (0.68) | -6.99 (0.92)
  Change at Week 9: number analyzed (Participants) | 146 | 74
  Change at Week 9 | -7.58 (0.71) | -8.14 (0.96)
  Change at Week 10: number analyzed (Participants) | 147 | 73
  Change at Week 10 | -7.71 (0.76) | -9.11 (1.04)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 6; Test type: Superiority; p = 0.2781, Mixed Models Analysis — The p-value was derived using MMRM method with treatment, study center, visit week, and treatment by visit week interaction as class effects, and week 5 value as covariate; Mean Difference (Final Values) = 0.81, 95% CI 2-sided [-0.66 to 2.28] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.4673, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-1.15 to 2.49] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 8; Test type: Superiority; p = 0.5719, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-1.54 to 2.79] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.6262, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-1.70 to 2.83] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 10; Test type: Superiority; p = 0.2638, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.40, 95% CI 2-sided [-1.06 to 3.87] — [estimate comment as in outcome 3, analysis 1]

7. Secondary Outcome: Change From Baseline (End of Phase A) in CAARS-O:SV Inattentive Symptoms Subscale Score (9 Items) to Each Time Point in Phase B
Description: The CAARS-O:SV is a 30 items scale with 3 subscales DSM-IV Inattentive Symptoms (9 items), DSM-IV Hyperactive/Impulsive Symptoms (9 items), and DSM-IV ADHD Index (12 items). The inattentive symptoms subscale (9 items) is scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) with total score ranging from 0 to 27, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)]; Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Change at Week 6 | -2.00 (0.32) | -2.43 (0.41)
  Change at Week 7: number analyzed (Participants) | 150 | 74
  Change at Week 7 | -2.94 (0.36) | -3.20 (0.48)
  Change at Week 8: number analyzed (Participants) | 150 | 74
  Change at Week 8 | -3.14 (0.40) | -3.42 (0.54)
  Change at Week 9: number analyzed (Participants) | 146 | 74
  Change at Week 9 | -3.74 (0.42) | -4.04 (0.57)
  Change at Week 10: number analyzed (Participants) | 147 | 73
  Change at Week 10 | -3.95 (0.45) | -4.85 (0.62)
  Change at Week 11: number analyzed (Participants) | 147 | 69
  Change at Week 11 | -4.58 (0.44) | -4.86 (0.60)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 6; Test type: Superiority; p = 0.3804, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.52 to 1.37] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.6422, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.86 to 1.39] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 8; Test type: Superiority; p = 0.6707, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-1.00 to 1.55] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.6638, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-1.04 to 1.64] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 10; Test type: Superiority; p = 0.2252, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [-0.56 to 2.36] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 11; Test type: Superiority; p = 0.6970, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-1.14 to 1.70] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: Change From Baseline (End of Phase A) in CAARS-O:SV Hyperactive/Impulsive Symptoms Subscale Score (9 Items) to Each Time Point in Phase B
Description: The CAARS-O:SV is a 30 items scale with 3 subscales DSM-IV Inattentive Symptoms (9 items), DSM-IV Hyperactive/Impulsive Symptoms (9 items), and DSM-IV ADHD Index (12 items). The hyperactive/impulsive Symptoms Subscale is (9 items) scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) with total score ranging from 0 to 27, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)]; Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Change at Week 6 | -1.88 (0.29) | -2.11 (0.38)
  Change at Week 7: number analyzed (Participants) | 150 | 74
  Change at Week 7 | -2.66 (0.32) | -2.94 (0.43)
  Change at Week 8: number analyzed (Participants) | 150 | 74
  Change at Week 8 | -3.29 (0.36) | -3.48 (0.49)
  Change at Week 9: number analyzed (Participants) | 146 | 74
  Change at Week 9 | -3.90 (0.39) | -4.01 (0.53)
  Change at Week 10: number analyzed (Participants) | 147 | 73
  Change at Week 10 | -3.83 (0.41) | -4.17 (0.55)
  Change at Week 11: number analyzed (Participants) | 147 | 69
  Change at Week 11 | -4.51 (0.42) | -4.80 (0.58)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 6; Test type: Superiority; p = 0.6008, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.64 to 1.11] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.5859, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.72 to 1.27] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 8; Test type: Superiority; p = 0.7406, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [-0.96 to 1.34] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.8568, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-1.14 to 1.37] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 10; Test type: Superiority; p = 0.6044, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.96 to 1.64] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 11; Test type: Superiority; p = 0.6772, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-1.08 to 1.66] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Change From Baseline (End of Phase A) in CAARS-O:SV ADHD Index Score (12 Items) to Each Time Point in Phase B
Description: The CAARS-S:SV is a 30 items scale with 3 subscales inattention (9 items), hyperactivity-impulsivity (9 items), and ADHD index (12 items). The ADHD index score (12 items) is scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) with total score ranging from 0 to 36, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)]; Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Change at Week 6 | -2.06 (0.34) | -2.20 (0.44)
  Change at Week 7: number analyzed (Participants) | 150 | 74
  Change at Week 7 | -3.47 (0.41) | -3.38 (0.55)
  Change at Week 8: number analyzed (Participants) | 150 | 74
  Change at Week 8 | -4.01 (0.44) | -3.80 (0.59)
  Change at Week 9: number analyzed (Participants) | 146 | 74
  Change at Week 9 | -4.32 (0.46) | -4.78 (0.62)
  Change at Week 10: number analyzed (Participants) | 147 | 73
  Change at Week 10 | -4.65 (0.47) | -5.23 (0.64)
  Change at Week 11: number analyzed (Participants) | 147 | 69
  Change at Week 11 | -5.60 (0.48) | -5.94 (0.66)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 6; Test type: Superiority; p = 0.7881, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.87 to 1.15] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.8841, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1.38 to 1.19] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 8; Test type: Superiority; p = 0.7589, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-1.61 to 1.17] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.5375, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-1.01 to 1.93] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 10; Test type: Superiority; p = 0.4456, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-0.92 to 2.08] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 11; Test type: Superiority; p = 0.6670, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-1.21 to 1.89] — [estimate comment as in outcome 3, analysis 1]

10. Secondary Outcome: Change From Baseline (End of Phase A) to Weeks 7 and 9 in ISI Total Score
Description: as for outcome 3
Time Frame: Baseline [end of Phase A (Week 5)]; Weeks 7 and 9
Population: Efficacy Sample=participants in Randomized Sample who had Baseline value for Phase B (ie Week 5) and at least one post-randomization efficacy evaluation for CAARS-O:SV ADHD symptoms Total Score (18 items) in Phase B. As prespecified in protocol, SAP data is reported only for Phase B participants. Overall number of participants=number of participants with data available for analyses at Baseline. Number analyzed=number of participants with data available for analyses at given timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 150 | 77
score on a scale
  Change at Week 7: number analyzed (Participants) | 148 | 74
  Change at Week 7 | -0.81 (0.33) | -0.83 (0.44)
  Change at Week 9: number analyzed (Participants) | 145 | 71
  Change at Week 9 | -0.99 (0.37) | -1.48 (0.49)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.9708, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.97 to 1.01] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.3970, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-0.65 to 1.63] — [estimate comment as in outcome 3, analysis 1]

11. Secondary Outcome: Percentage of Participants With Categorical Change in Sleep Improvement Measured by Individual Scores for Items 1, 2, and 3 of the ISI at End of Phase B
Description: The ISI is self-report instrument that has been validated specifically for measuring the perceived severity of insomnia. The scale was composed of a total of 7 items based on self-report questionnaire based on several indicators assessing the perceived severity. difficulties initiating sleep, staying asleep, and early morning awakenings, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item was rated on a scale from 0 (none) to 4 (higher score indicating greater impairment/concern). A negative change from Baseline indicates improvement. The Cochran-Mantel-Haenszel model was used for analysis.
Time Frame: Baseline [(end of Phase A (Week 5)] to Weeks 7, 9 and 11
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
percentage of participants
  Difficulty Falling Asleep: Week 7: number analyzed (Participants) | 149 | 74
  Difficulty Falling Asleep: Week 7 | 33.6 | 32.4
  Difficulty Falling Asleep: Week 9: number analyzed (Participants) | 150 | 77
  Difficulty Falling Asleep: Week 9 | 33.3 | 37.7
  Difficulty Falling Asleep: Week 11: number analyzed (Participants) | 150 | 77
  Difficulty Falling Asleep: Week 11 | 35.3 | 39.0
  Difficulty Staying Asleep: Week 7: number analyzed (Participants) | 149 | 74
  Difficulty Staying Asleep: Week 7 | 26.8 | 35.1
  Difficulty Staying Asleep: Week 9: number analyzed (Participants) | 150 | 77
  Difficulty Staying Asleep: Week 9 | 25.3 | 33.8
  Difficulty Staying Asleep: Week 11: number analyzed (Participants) | 150 | 77
  Difficulty Staying Asleep: Week 11 | 24.7 | 37.7
  Waking Up Too Early: Week 7: number analyzed (Participants) | 149 | 74
  Waking Up Too Early: Week 7 | 28.2 | 25.7
  Waking Up Too Early: Week 9: number analyzed (Participants) | 150 | 77
  Waking Up Too Early: Week 9 | 30.7 | 26.0
  Waking Up Too Early: Week 11: number analyzed (Participants) | 150 | 77
  Waking Up Too Early: Week 11 | 29.3 | 28.6
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Difficulty Falling Asleep: Week 7; Test type: Superiority; p = 0.9568, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.68 to 1.50] — The difference between LS means derived from the Cochran-Mantel-Haenszel (CMH) model. This comparison was tested for statistical significance at a 0.05 (two-sided) significance level
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Difficulty Falling Asleep: Week 9; Test type: Superiority; p = 0.6308, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.63 to 1.31] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Difficulty Falling Asleep: Week 11; Test type: Superiority; p = 0.6698, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.64 to 1.32] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Difficulty Staying Asleep: Week 7; Test type: Superiority; p = 0.2012, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.76, 95% CI 2-sided [0.50 to 1.15] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Difficulty Staying Asleep: Week 9; Test type: Superiority; p = 0.2365, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.52 to 1.16] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Difficulty Staying Asleep: Week 11; Test type: Superiority; p = 0.0312, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.65, 95% CI 2-sided [0.44 to 0.96] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 7: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Waking Up Too Early: Week 7; Test type: Superiority; p = 0.6408, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.69 to 1.81] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 8: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Waking Up Too Early: Week 9; Test type: Superiority; p = 0.3467, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.24, 95% CI 2-sided [0.79 to 1.96] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 9: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Waking Up Too Early: Week 11; Test type: Superiority; p = 0.9437, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.65 to 1.59] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Change From Baseline (End of Phase A) in Conners' Adult ADHD Rating Scale-Self-Report: Screening Version (CAARS-S:SV) ADHD Symptoms Total Score (18 Items) to Each Timepoint in Phase B
Description: The CAARS-S:SV is a self-reported 30 items scale with 3 subscales inattention (9 items), hyperactivity-impulsivity (9 items), and ADHD index (12 items). Total ADHD Symptoms Score (18 items) consisted of the combined score for the Inattentive Symptoms and Hyperactive/Impulsive Symptoms subscales and is scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) for total score ranging from of 0 to 54, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)]; Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Change at Week 6 | -1.75 (0.58) | -2.16 (0.75)
  Change at Week 7: number analyzed (Participants) | 150 | 74
  Change at Week 7 | -3.01 (0.65) | -3.47 (0.87)
  Change at Week 8: number analyzed (Participants) | 150 | 74
  Change at Week 8 | -4.15 (0.68) | -4.08 (0.92)
  Change at Week 9: number analyzed (Participants) | 146 | 74
  Change at Week 9 | -4.24 (0.73) | -5.23 (0.99)
  Change at Week 10: number analyzed (Participants) | 147 | 73
  Change at Week 10 | -4.63 (0.77) | -6.11 (1.04)
  Change at Week 11: number analyzed (Participants) | 147 | 69
  Change at Week 11 | -5.38 (0.78) | -6.33 (1.07)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 6; Test type: Superiority; p = 0.6357, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-1.30 to 2.12] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.6536, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [-1.56 to 2.48] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 8; Test type: Superiority; p = 0.9475, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-2.20 to 2.06] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.3973, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.99, 95% CI 2-sided [-1.31 to 3.29] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 10; Test type: Superiority; p = 0.2336, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.47, 95% CI 2-sided [-0.96 to 3.91] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 11; Test type: Superiority; p = 0.4553, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.95, 95% CI 2-sided [-1.55 to 3.44] — [estimate comment as in outcome 3, analysis 1]

13. Secondary Outcome: Change From Baseline (End of Phase A) in CAARS-S:SV Inattentive Symptoms Subscale Score (9 Items) to Each Timepoint in Phase B
Description: The CAARS-S:SV is a self-reported 30 items scale with 3 subscales inattention (9 items), hyperactivity-impulsivity (9 items), and ADHD index (12 items). The Inattentive Symptoms Subscale is (9 items) scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) with total score ranging from 0 to 27, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)]; Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Change at Week 6 | -0.87 (0.33) | -1.16 (0.43)
  Change at Week 7: number analyzed (Participants) | 150 | 74
  Change at Week 7 | -1.64 (0.37) | -1.62 (0.49)
  Change at Week 8: number analyzed (Participants) | 150 | 74
  Change at Week 8 | -2.08 (0.40) | -1.93 (0.54)
  Change at Week 9: number analyzed (Participants) | 146 | 74
  Change at Week 9 | -2.08 (0.42) | -2.42 (0.56)
  Change at Week 10: number analyzed (Participants) | 147 | 73
  Change at Week 10 | -2.43 (0.43) | -2.84 (0.58)
  Change at Week 11: number analyzed (Participants) | 147 | 69
  Change at Week 11 | -2.54 (0.43) | -3.10 (0.59)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 6; Test type: Superiority; p = 0.5647, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.70 to 1.27] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.9739, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-1.15 to 1.12] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 8; Test type: Superiority; p = 0.8077, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-1.40 to 1.09] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.6119, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.34, 95% CI 2-sided [-0.98 to 1.65] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 10; Test type: Superiority; p = 0.5513, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-0.94 to 1.76] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 11; Test type: Superiority; p = 0.4185, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-0.81 to 1.95] — [estimate comment as in outcome 3, analysis 1]

14. Secondary Outcome: Change From Baseline (End of Phase A) in CAARS-S:SV Hyperactive/Impulsive Symptoms Subscale Score (9 Items) to Each Timepoint in Phase B
Description: The CAARS-S:SV is a 30 items scale with 3 subscales inattention (9 items), hyperactivity-impulsivity (9 items), and ADHD index (12 items). The Hyperactive/Impulsive Symptoms Subscale is (9 items) scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) with total score ranging from 0 to 27, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)]; Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Change at Week 6 | -0.91 (0.32) | -1.06 (0.41)
  Change at Week 7: number analyzed (Participants) | 150 | 74
  Change at Week 7 | -1.38 (0.35) | -1.88 (0.47)
  Change at Week 8: number analyzed (Participants) | 150 | 74
  Change at Week 8 | -2.09 (0.36) | -2.20 (0.47)
  Change at Week 9: number analyzed (Participants) | 146 | 74
  Change at Week 9 | -2.18 (0.39) | -2.87 (0.52)
  Change at Week 10: number analyzed (Participants) | 147 | 73
  Change at Week 10 | -2.21 (0.41) | -3.33 (0.55)
  Change at Week 11: number analyzed (Participants) | 147 | 69
  Change at Week 11 | -2.86 (0.42) | -3.31 (0.57)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 6; Test type: Superiority; p = 0.7556, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.80 to 1.09] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.3710, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-0.60 to 1.59] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 8; Test type: Superiority; p = 0.8464, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.99 to 1.21] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.2664, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [-0.53 to 1.91] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 10; Test type: Superiority; p = 0.0876, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 1.13, 95% CI 2-sided [-0.17 to 2.42] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 11; Test type: Superiority; p = 0.5119, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.89 to 1.77] — [estimate comment as in outcome 3, analysis 1]

15. Secondary Outcome: Change From Baseline (End of Phase A) in CAARS-S:SV ADHD Index Score (12 Items) to Each Timepoint in Phase B
Description: The CAARS-S:SV is a 30 items scale with 3 subscales inattention (9 items), hyperactivity-impulsivity (9 items), and ADHD index (12 items). The ADHD Index Subscale is (12 items) scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) with total score ranging from 0 to 36, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)]; Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Change at Week 6 | -1.09 (0.37) | -1.16 (0.48)
  Change at Week 7: number analyzed (Participants) | 150 | 74
  Change at Week 7 | -1.86 (0.42) | -2.13 (0.55)
  Change at Week 8: number analyzed (Participants) | 150 | 74
  Change at Week 8 | -2.69 (0.44) | -2.43 (0.59)
  Change at Week 9: number analyzed (Participants) | 146 | 74
  Change at Week 9 | -3.07 (0.46) | -3.00 (0.61)
  Change at Week 10: number analyzed (Participants) | 147 | 73
  Change at Week 10 | -3.42 (0.47) | -3.56 (0.63)
  Change at Week 11: number analyzed (Participants) | 147 | 69
  Change at Week 11 | -4.05 (0.48) | -3.90 (0.65)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 6; Test type: Superiority; p = 0.8986, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-1.03 to 1.18] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.6850, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-1.02 to 1.55] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 8; Test type: Superiority; p = 0.7108, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-1.61 to 1.10] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.9236, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-1.50 to 1.36] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 10; Test type: Superiority; p = 0.8576, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-1.35 to 1.61] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 11; Test type: Superiority; p = 0.8483, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-1.67 to 1.37] — [estimate comment as in outcome 3, analysis 1]

16. Secondary Outcome: Change From Baseline (End of Phase A) in Clinical Global Impression - Severity of Illness Scale (CGI-S) Score to Each Timepoint in Phase B
Description: The CGI-S is performed to rate the severity of a participant's condition on an 8-point scale ranging from 0 to 7 where 0=not assessed, 1=normal, not at all ill, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7 = among the most extremely ill participants. A negative change from Baseline indicates improvement. The MMRM model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)]; Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Change at Week 6 | -0.75 (0.06) | -0.71 (0.08)
  Change at Week 7: number analyzed (Participants) | 150 | 74
  Change at Week 7 | -0.92 (0.07) | -0.88 (0.09)
  Change at Week 8: number analyzed (Participants) | 150 | 74
  Change at Week 8 | -1.03 (0.07) | -0.97 (0.10)
  Change at Week 9: number analyzed (Participants) | 146 | 74
  Change at Week 9 | -1.16 (0.08) | -1.10 (0.11)
  Change at Week 10: number analyzed (Participants) | 147 | 73
  Change at Week 10 | -1.17 (0.08) | -1.28 (0.11)
  Change at Week 11: number analyzed (Participants) | 147 | 69
  Change at Week 11 | -1.31 (0.09) | -1.37 (0.12)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 6; Test type: Superiority; p = 0.6976, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.22 to 0.15] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 7; Test type: Superiority; p = 0.6986, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.25 to 0.17] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 8; Test type: Superiority; p = 0.6507, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.30 to 0.19] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 9; Test type: Superiority; p = 0.6550, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.32 to 0.20] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 10; Test type: Superiority; p = 0.3959, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.15 to 0.38] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Change at Week 11; Test type: Superiority; p = 0.6763, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.23 to 0.35] — [estimate comment as in outcome 3, analysis 1]

17. Secondary Outcome: Change From Baseline (End of Phase A) in the SWM Strategy 6-8 Boxes Test Score as Measured by CANTAB to End of Phase B
Description: The SWM test assesses the cognitive domain of executive function (high-level thinking and decision making). SWM task was SWM Strategy 6-8 Boxes, in which the total number of distinct boxes used by the participant to begin a new search for a token within the same problem was measured for the 6- and 8-box stages. The SWM strategy index of executive function represented the number of times a participant began a search with a different box. Participant was asked to find tokens in on-screen boxes and move them. Difficulty ranged from 4 to 8 box assessments. Strategy score was the number of unique boxes the participant searched in 6 and 8 box trials. 6 box trial scores ranged from 1 (1 box searched for all 6 tokens) to 6 (6 boxes searched for 6 tokens). 8 box trial score ranged from 1 (1 box searched) to 8 (8 boxes searched for 8 tokens). Total of the 2 trial scores ranged from 2 to 14. A lower score reflects better performance. The ANCOVA method was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 145 | 72
score on a scale | 0.15 (0.21) | -0.12 (0.28)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.4089, ANCOVA — The p-value was derived from ANCOVA model, with treatment and study center as main effects and week 5 value as covariate, is used for change from week 5 comparisons; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.37 to 0.91] — [estimate comment as in outcome 2, analysis 1]

18. Secondary Outcome: Change From Baseline (End of Phase A) in the SWM Within Errors 4-8 Boxes Test Score as Measured by CANTAB to End of Phase B
Description: Assessments were performed with CANTAB. SWM test assesses cognitive domain of executive function (high-level thinking and decision making). Participants search for colored tokens hidden inside boxes on screen by touching them. Critical instruction is that once a token has been found inside a box, there was never be a token hidden inside that box again, so participants must not return to a box where a token has been found. Within Errors 4-8 Boxes, which measured number of times a participant revisited a box that had already been found to be empty during the same search. Value was reported as total number of errors for 4-, 6-, and 8-box stages. Observed range for Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant is -8.00 to 6.00 (change from baseline) and for Phase B (Double-blind Randomization Phase): Placebo + Stimulant is -10.0 to 23.00 (change from baseline). A lower score reflects better performance. LOCF method was used to impute missing data.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 145 | 72
score on a scale | 0.00 (0.16) | 0.30 (0.22)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority or Other; p = 0.2331, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.80 to 0.20] — Week 11 data is included here. The planned sample size of 225 participants (150 in brexipiprazole arm and 75 in the placebo arm) yielded at least 80% power to detect effects at a 2-tailed significance level of 0.05 using a two-sided z-test

19. Secondary Outcome: Change From Baseline (End of Phase A) in the Rapid Visual Information Processing (RVP) A Prime Test Score as Measured by CANTAB to End of Phase B
Description: Assessments were performed with the CANTAB. The RVP task tested continuous performance and visual sustained attention. In the center of the computer screen, digits from 2 to 9 appear inside a white box in pseudorandom order at a rate of 100 digits per minute. Participants must touch the press pad when they detect a series of target digit sequences (eg, 2-4-6, 4-6-8, 3-5-7) which appeared at a rate of 9 sequences every 100 numbers. Data from the RVP task were summarized in 3 ways: RVP A prime, RVP median response latency, and RVP total false alarms. RVP A prime was the signal detection measure of sensitivity to the target, regardless of response tendency (range 0.00 to 1.00; bad to good). In essence, this metric was a measure of how good the participant was at detecting target sequences. Higher scores indicated better performance. The ANCOVA method was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 145 | 72
score on a scale | 0.00 (0.00) | 0.01 (0.00)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.0670, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.01 to 0.00] — [estimate comment as in outcome 2, analysis 1]

20. Secondary Outcome: Change From Baseline (End of Phase A) in the RVP Median Response Latency Score as Measured by CANTAB to End of Phase B
Description: Assessments were performed with CANTAB. RVP task tested continuous performance and visual sustained attention. In the center of computer screen, digits from 2 to 9 appear inside white box in pseudorandom order at a rate of 100 digits per minute. Participants must touch press pad when they detect a series of target digit sequences (eg, 2-4-6, 4-6-8, 3-5-7) which appeared at a rate of 9 sequences every 100 numbers. Data from RVP task were summarized in 3 ways: RVP A prime, RVP median response latency, and RVP total false alarms. Median response latency was measured during the assessed part of test (7-minute continuous part of test after initial 2 minutes training phase). Observed range for Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant is -338 to 282.0 (change from baseline) and for Phase B (Double-blind Randomization Phase): Placebo + Stimulant is -134 to 235.0 (change from baseline). Lower scores indicate better performance. ANCOVA method was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 145 | 72
score on a scale | -17.1 (5.36) | -2.89 (7.10)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.0849, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = -14.3, 95% CI 2-sided [-30.5 to 1.98] — [estimate comment as in outcome 2, analysis 1]

21. Secondary Outcome: Change From Baseline (End of Phase A) in RVP Total False Alarms Score as Measured by CANTAB to End of Phase B
Description: RVP task tested continuous performance and visual sustained attention. In center of computer screen, digits from 2- 9 appear inside a white box in pseudorandom order at a rate of 100 digits per minute. Participants must touch press pad when they detect a series of target digit sequences (e.g., 2-4-6, 4-6-8, 3-5-7) which appeared at a rate of 9 sequences every 100 numbers. Data from RVP task were summarized in 3 ways: RVP A prime, RVP median response latency, and RVP total false alarms. False alarms were determined from number of times that participants responded outside response window of a target sequence during assessed part of test. Observed range for Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant is -26.0 to 13.00 (change from baseline) and for Phase B (Double-blind Randomization Phase): Placebo + Stimulant is -25.0 to 144.0 (change from baseline). Lower scores indicate better performance. ANCOVA model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 145 | 72
score on a scale | 0.12 (1.01) | 0.58 (1.34)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.7663, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-3.52 to 2.60] — [estimate comment as in outcome 2, analysis 1]

22. Secondary Outcome: Change From Baseline (End of Phase A) in the Stop Signal Task (SST) Stop Signal Reaction Time (SSRT) Score as Measured by CANTAB to End of Phase B
Description: In SST, an arrow pointing either left or right is displayed on computer screen. Participant responded to arrow by pressing corresponding button (i.e., left or right) on press pad. If an audio tone is presented when arrow is displayed, participant inhibited response. Proportion of successful stops, and median reaction time on Go trials was measured. SST SSRT was an estimate of length of time between go stimulus and stop stimulus at which participant was able to successfully inhibit response on 50% of trials and calculated from SST reaction time on Go trials measure and SST stop signal delay (SSD) 50% measure as [reaction time on Go trials] - [SSD (50%)], where SSD (50%) measure was calculated as arithmetic mean of measured SSD, or failed stop reaction time, from completed assessment stop trials. Observed change from baseline range for Phase B: Brexpiprazole + Stimulant: -204 to 237.0 and for Phase B: Placebo + Stimulant: -176 to 113.0. Lower scores indicate better performance.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 145 | 72
score on a scale | 13.41 (5.12) | -4.10 (6.92)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.0298, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = 17.51, 95% CI 2-sided [1.73 to 33.29] — [estimate comment as in outcome 2, analysis 1]

23. Secondary Outcome: Change From Baseline (End of Phase A) in the SST Proportion of Successful Stops Score as Measured by CANTAB to End of Phase B
Description: SST measures participants ability to inhibit a response. An arrow pointing either left or right is displayed on computer screen. Participant responded to arrow by pressing corresponding button (i.e., left or right) on press pad. If an audio tone is presented when arrow is displayed, participant inhibited his/her response. Proportion of successful stops, and median reaction time on Go trials was measured. The proportion of successful stops is calculated as the number of times that the participant stopped successfully, divided by the total number of stop signals. Observed range for Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant: -0.40 to 0.40 (change from baseline) and for Phase B (Double-blind Randomization Phase): Placebo + Stimulant: -0.38 to 0.38 (change from baseline). Higher scores indicate a positive outcome for proportion of successful stops.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 145 | 72
score on a scale | -0.01 (0.01) | 0.01 (0.01)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.2563, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.05 to 0.01] — [estimate comment as in outcome 2, analysis 1]

24. Secondary Outcome: Change From Baseline (End of Phase A) in SST Median Reaction Time Score on Go Trials as Measured by CANTAB to End of Phase B
Description: SST measures participants ability to inhibit a response. An arrow pointing either left or right is displayed on computer screen. Participant responded to arrow by pressing corresponding button (i.e., left or right) on press pad. If an audio tone is presented when arrow is displayed, participant inhibited his/her response. Proportion of successful stops, and median reaction time on Go trials was measured. The median reaction time on Go trials is the median of the reaction time assessed on Go trials to which the participant responded correctly. Observed range for Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant: -277 to 266.0 (change from baseline) and for Phase B (Double-blind Randomization Phase): Placebo + Stimulant: -462 to 358.0 (change from baseline). Lower scores indicate better performance.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 145 | 72
score on a scale | -6.70 (8.39) | -1.03 (11.2)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.6644, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = -5.67, 95% CI 2-sided [-31.4 to 20.06] — [estimate comment as in outcome 2, analysis 1]

25. Secondary Outcome: Change From Baseline (End of Phase A) in WRAADDS Attention + Organization Subscale Score to End of Phase B
Description: WRAADDS is used to measure the severity of symptoms in adults with ADHD. This structured interview consists of 28 items in 7 psychopathologic domains, which were rated by a clinical expert on a 0 to 2-point Likert scale. The psychopathologic 7 domains are inattention (6 items), impulsivity (3 items), and hyperactivity (3 items), disorganization (5 items), temper (3 items), affective lability (4 items), and emotional over-reactivity (4 items). The scale rated individual items from 0 to 2 (0=not present, 1=mild, 2=clearly present). The score for attention + organization subscale score ranges from 0-22, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The ANCOVA method was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 150 | 74
score on a scale | -1.47 (0.17) | -1.42 (0.22)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.8418, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.56 to 0.45] — [estimate comment as in outcome 2, analysis 1]

26. Secondary Outcome: Change From End of Phase A (Week 5 Visit) to End of Phase B (Week 11 Visit) in WRAADDS Hyperactivity + Impulsivity Subscale Score to End of Phase B
Description: WRAADDS is used to measure the severity of symptoms in adults with ADHD. This structured interview consists of 28 items in 7 psychopathologic domains, which were rated by a clinical expert on a 0 to 2-point Likert scale. The psychopathologic 7 domains are inattention (6 items), impulsivity (3 items), and hyperactivity (3 items), disorganization (5 items), temper (3 items), affective lability (4 items), and emotional over-reactivity (4 items). The scale rated individual items from 0 to 2 (0=not present, 1=mild, 2=clearly present). The score for hyperactivity + impulsivity subscale score ranges from 0-12, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The ANCOVA model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 150 | 74
score on a scale | -1.27 (0.14) | -1.01 (0.19)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.2513, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.69 to 0.18] — [estimate comment as in outcome 2, analysis 1]

27. Secondary Outcome: Change From Baseline (End of Phase A) in WRAADDS Temper + Mood Lability + Emotional Over-reactivity Subscale Score to End of Phase B
Description: WRAADDS is used to measure the severity of symptoms in adults with ADHD. This structured interview consists of 28 items in 7 psychopathologic domains, which were rated by a clinical expert on a 0 to 2-point Likert scale. The psychopathologic 7 domains are inattention (6 items), impulsivity (3 items), and hyperactivity (3 items), disorganization (5 items), temper (3 items), affective lability (4 items), and emotional over-reactivity (4 items). The scale rated individual items from 0 to 2 (0=not present, 1=mild, 2=clearly present). The score for temper + mood Lability + emotional over-reactivity subscale score ranges from 0-22, higher scores indicate worsening of symptoms. A negative change from Baseline indicates improvement. The ANCOVA model was used for analysis.
Time Frame: Baseline [end of Phase A (Week 5)] to Week 11
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 150 | 74
score on a scale | -1.24 (0.20) | -1.35 (0.26)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Test type: Superiority; p = 0.7037, ANCOVA — [p-value comment as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.48 to 0.71] — [estimate comment as in outcome 2, analysis 1]

28. Secondary Outcome: Mean CGI-I Score at Each Timepoint in Phase B
Description: The CGI-I permits a global evaluation of the participant's improvement over time. The CGI-I is a 8-point scale ranging from 0 to 7 where 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse and 7=very much worse. The CGI-I is completed by the clinician and assesses the participant's improvement relative to the symptoms at Baseline. The Cochran-Mantel-Haenszel model was used for analysis.
Time Frame: Weeks 6, 7, 8, 9, 10 and 11
Population: Efficacy Sample consisted of participants in the Randomized Sample who had a Baseline value for Phase B (ie, Week 5) and at least one post-randomization efficacy evaluation for CAARS-O:SV ADHD symptoms Total Score (18 items) in Phase B. As pre-specified in the protocol and SAP the data is reported only for Phase B participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
score on a scale
  Week 6 | 3.19 (0.81) | 3.12 (0.77)
  Week 7 | 3.04 (0.88) | 3.08 (0.80)
  Week 8 | 2.93 (0.96) | 2.88 (1.01)
  Week 9 | 2.82 (1.02) | 2.81 (1.03)
  Week 10 | 2.80 (0.99) | 2.76 (1.07)
  Week 11 | 2.68 (1.06) | 2.69 (1.17)
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 6; Test type: Superiority; p = 0.7572, Cochran-Mantel-Haenszel — The p-value was derived from CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.17 to 0.23] — The difference between LS means derived from the CMH model. This comparison was tested for statistical significance at a 0.05 (two-sided) significance level
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 7; Test type: Superiority; p = 0.6132, Cochran-Mantel-Haenszel — The p-value was derived from CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.28 to 0.17] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 8; Test type: Superiority; p = 0.9312, Cochran-Mantel-Haenszel — The p-value was derived from CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.25 to 0.27] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 9; Test type: Superiority; p = 0.8073, Cochran-Mantel-Haenszel — The p-value was derived from CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.30 to 0.24] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 10; Test type: Superiority; p = 0.9168, Cochran-Mantel-Haenszel — The p-value was derived from CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.26 to 0.29] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 11; Test type: Superiority; p = 0.7432, Cochran-Mantel-Haenszel — The p-value was derived from CMH row mean scores differ test controlling for study center; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.34 to 0.25] — [estimate comment as in outcome 28, analysis 1]

29. Secondary Outcome: Percentage of Participants With CAARS-O:SV ADHD Symptoms Response Rate in Phase B
Description: Response was defined as ≥ 30% reduction in CAARS-O:SV ADHD Symptoms Total Score (18 items) from end of Phase A (Week 5 visit). An 18-item ADHD Symptoms Total Score consisted of the combined score for the Inattentive Symptoms and Hyperactive/Impulsive Symptoms subscales. The CAARS-O:SV was designed to measure a cross-section of ADHD-related symptoms and behaviors in adults using observer and self-report scales. Total ADHD Symptoms Score (18 items) consisted of the combined score for the inattentive symptoms and hyperactive/impulsive symptoms subscales and is scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) for a total score ranging from of 0 to 54, higher scores indicate worsening of symptoms.
Time Frame: Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
percentage of participants
  Week 6 | 15.0 | 12.8
  Week 7 | 24.2 | 24.4
  Week 8 | 28.8 | 33.3
  Week 9 | 35.9 | 41.0
  Week 10 | 37.9 | 44.9
  Week 11 | 45.1 | 50.0
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 6; Test type: Superiority; p = 0.6014, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.20, 95% CI 2-sided [0.60 to 2.42] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 7; Test type: Superiority; p = 0.9225, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.64 to 1.63] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 8; Test type: Superiority; p = 0.4803, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.58 to 1.30] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 9; Test type: Superiority; p = 0.5876, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.65 to 1.27] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 10; Test type: Superiority; p = 0.3727, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.64 to 1.18] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 11; Test type: Superiority; p = 0.6265, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.71 to 1.23] — [estimate comment as in outcome 28, analysis 1]

30. Secondary Outcome: Percentage of Participants With CAARS-O:SV ADHD Symptoms Remission Rate in Phase B
Description: Remission was defined as CAARS-O:SV ADHD Symptoms Total Score (18 items) of ≤ 18 and a ≥ 30% reduction in CAARS-O:SV ADHD Symptoms Total Score (18 items) from end of Phase A (Week 5 visit). An 18-item ADHD Symptoms Total Score consisted of the combined score for the Inattentive Symptoms and Hyperactive/Impulsive Symptoms subscales. The CAARS-O:SV was designed to measure a cross-section of ADHD-related symptoms and behaviors in adults using observer and self-report scales. Total ADHD Symptoms Score (18 items) consisted of the combined score for the inattentive symptoms and hyperactive/impulsive symptoms subscales and is scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) for a total score ranging from of 0 to 54, higher scores indicate worsening of symptoms. The Cochran-Mantel-Haenszel model was used for analysis.
Time Frame: Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
percentage of participants
  Week 6 | 7.19 | 6.41
  Week 7 | 12.4 | 12.8
  Week 8 | 19.0 | 19.2
  Week 9 | 20.9 | 23.1
  Week 10 | 25.5 | 28.2
  Week 11 | 27.5 | 33.3
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 6; Test type: Superiority; p = 0.8586, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.40 to 3.03] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 7; Test type: Superiority; p = 0.8984, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.46 to 1.99] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 8; Test type: Superiority; p = 0.9778, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.57 to 1.74] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 9; Test type: Superiority; p = 0.7315, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.56 to 1.50] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 10; Test type: Superiority; p = 0.6518, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.57 to 1.42] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 11; Test type: Superiority; p = 0.3472, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.55 to 1.23] — [estimate comment as in outcome 28, analysis 1]

31. Secondary Outcome: Percentage of Participants With CAARS-S:SV ADHD Symptoms Response Rate in Phase B
Description: Response was defined as ≥ 30% reduction in CAARS-S:SV ADHD Symptoms Total Score (18 items) from end of Phase A (Week 5 visit). The CAARS-S:SV is a 30 items scale with 3 subscales inattention (9 items), hyperactivity-impulsivity (9 items), and ADHD index (12 items). Total ADHD Symptoms Score (18 items) consisted of the combined score for the Inattentive Symptoms and Hyperactive/Impulsive Symptoms subscales is scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) for total score ranging from of 0 to 54, higher scores indicate worsening of symptoms. The Cochran-Mantel-Haenszel model was used for analysis.
Time Frame: Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
percentage of participants
  Week 6 | 11.8 | 12.8
  Week 7 | 18.3 | 15.4
  Week 8 | 21.6 | 21.8
  Week 9 | 29.4 | 29.5
  Week 10 | 25.5 | 32.1
  Week 11 | 31.4 | 37.2
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 6; Test type: Superiority; p = 0.9577, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.44 to 2.16] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 7; Test type: Superiority; p = 0.5864, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.19, 95% CI 2-sided [0.63 to 2.27] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 8; Test type: Superiority; p = 0.8723, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.57 to 1.60] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 9; Test type: Superiority; p = 0.9872, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.65 to 1.52] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 10; Test type: Superiority; p = 0.3171, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.52 to 1.23] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 11; Test type: Superiority; p = 0.4782, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.60 to 1.27] — [estimate comment as in outcome 28, analysis 1]

32. Secondary Outcome: Percentage of Participants With CAARS-S:SV ADHD Symptoms Remission Rate in Phase B
Description: Remission was defined as CAARS-S:SV ADHD Symptoms Total Score (18 items) of ≤ 18 and a ≥ 30% reduction in CAARS-S:SV ADHD Symptoms Total Score (18 items) from end of Phase A (Week 5 visit). The CAARS-S:SV is a 30 items scale with 3 subscales inattention (9 items), hyperactivity-impulsivity (9 items), and ADHD index (12 items). Total ADHD Symptoms Score (18 items) consisted of the combined score for the Inattentive Symptoms and Hyperactive/Impulsive Symptoms subscales is scored on a 4-point scale from 0 (not at all; never) to 3 (very much, very frequently) for total score ranging from of 0 to 54, higher scores indicate worsening of symptoms. The Cochran-Mantel-Haenszel model was used for analysis.
Time Frame: Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
percentage of participants
  Week 6 | 8.50 | 7.69
  Week 7 | 12.4 | 12.8
  Week 8 | 15.7 | 15.4
  Week 9 | 20.9 | 20.5
  Week 10 | 20.9 | 19.2
  Week 11 | 24.2 | 25.6
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 6; Test type: Superiority; p = 0.7232, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.19, 95% CI 2-sided [0.45 to 3.19] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 7; Test type: Superiority; p = 0.9860, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.46 to 2.13] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 8; Test type: Superiority; p = 0.9858, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.52 to 1.95] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 9; Test type: Superiority; p = 0.9466, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.58 to 1.78] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 10; Test type: Superiority; p = 0.6962, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.12, 95% CI 2-sided [0.63 to 2.00] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 11; Test type: Superiority; p = 0.7637, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.57 to 1.51] — [estimate comment as in outcome 28, analysis 1]

33. Secondary Outcome: Percentage of Participants With CGI-I Response Rate in Phase B
Description: Response was defined as a CGI-I score of 1 or 2 (very much improved or much improved). The CGI-I permits a global evaluation of the participant's improvement over time. The CGI-I is a 8-point scale ranging from 0 to 7 where 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse and 7=very much worse. The Cochran-Mantel-Haenszel model was used for analysis.
Time Frame: Weeks 6, 7, 8, 9, 10 and 11
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant
Number analyzed (Participants) | 153 | 78
percentage of participants
  Week 6 | 18.3 | 15.4
  Week 7 | 23.5 | 17.9
  Week 8 | 31.4 | 30.8
  Week 9 | 37.9 | 41.0
  Week 10 | 40.5 | 39.7
  Week 11 | 44.4 | 44.9
Statistical Analysis 1: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 6; Test type: Superiority; p = 0.3631, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.30, 95% CI 2-sided [0.73 to 2.33] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 2: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 7; Test type: Superiority; p = 0.2786, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.35, 95% CI 2-sided [0.78 to 2.35] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 3: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 8; Test type: Superiority; p = 0.7062, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.72 to 1.62] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 4: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 9; Test type: Superiority; p = 0.7844, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.67 to 1.35] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 5: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 10; Test type: Superiority; p = 0.6940, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.77 to 1.48] — [estimate comment as in outcome 28, analysis 1]
Statistical Analysis 6: Comparison: Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant vs Phase B (Double-blind Randomization Phase): Placebo + Stimulant; Week 11; Test type: Superiority; p = 0.8697, Cochran-Mantel-Haenszel — The p-value was derived from CMH general association test controlling for study center; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.76 to 1.39] — [estimate comment as in outcome 28, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after last dose of study drug (Up to approximately Week 15)
Description: Safety Sample consisted of randomized participants who received at least one dose of double-blind IMP as indicated on the dosing record. As pre-specified in the protocol the data for adverse events is presented in Part A, Part B and Part A+ as per the dose received.
Groups:
- Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant: Participants with incomplete response (with a > 0% and < 30% reduction in ADHD Symptoms Total Score {18 items} between the Baseline of Phase A and the end of prospective treatment {Week 5} as measured by the CAARS-O:SV {Conners' Adult ADHD Rating Scale-Observer: Screening Version}, and a CAARS-O:SV ADHD Symptoms Total Score {18 items} of ≥ 24 at Week 5, and a CGI-I score of 3 or 4 at Week 5) at the end of Phase A (Week 5), received Brexpiprazole 2mg tablet along with stimulant determined by the investigator, once daily for 6 weeks (up to Week 11).
Arm/Group | Phase A (Single-blind Prospective Treatment Phase): Placebo + Stimulant | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant | Phase B (Double-blind Randomization Phase): Placebo + Stimulant | Phase A+ (Single-blind Phase A Responders and Non-responders): Placebo + Stimulant
All-Cause Mortality (participants affected / at risk) | 0/733 | 0/155 | 0/80 | 0/339
Serious Adverse Events (participants affected / at risk) | 0/733 | 0/155 | 2/80 | 0/339
Other Adverse Events (participants affected / at risk) | 440/733 | 32/155 | 25/80 | 17/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase A (Single-blind Prospective Treatment Phase): Placebo + Stimulant (N=733) | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant (N=155) | Phase B (Double-blind Randomization Phase): Placebo + Stimulant (N=80) | Phase A+ (Single-blind Phase A Responders and Non-responders): Placebo + Stimulant (N=339)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase A (Single-blind Prospective Treatment Phase): Placebo + Stimulant (N=733) | Phase B (Double-blind Randomization Phase): Brexpiprazole + Stimulant (N=155) | Phase B (Double-blind Randomization Phase): Placebo + Stimulant (N=80) | Phase A+ (Single-blind Phase A Responders and Non-responders): Placebo + Stimulant (N=339)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 5 | 0
Weight decreased (Investigations) | 47 | 5 | 6 | 0
Headache (Nervous system disorders) | 128 | 11 | 10 | 0
Insomnia (Psychiatric disorders) | 0 | 13 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 113 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 51 | 0 | 0 | 0
Irritability (General disorders) | 57 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 155 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 44 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 43 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 85 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.